CLINICAL TRIAL: NCT06332729
Title: Effect of Universal Exercise Unit Versus Functional Electrical Stimulation On Genu Recurvatum In Diplegic Cerebral Palsy Children
Brief Title: Universal Exercise Unit Versus Functional Electrical Stimulation On Genu Recurvatum In Diplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahmoud Reda Elsharkawy (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Reda Elsharkawy, Demonstrator of pediatric department of physical therapy at Alsalam university, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EG,KFS,lab reserach 6
Record Dates: First submitted 2024-03-15; First posted 2024-03-27 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; universal exercise unit; functional electrical stimulation; diplegic; genu recurvatum
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- effect of universal exercis unit on genu recurvatum in diplegic cerbral palsy children (Active Comparator): Universal exercise unit (UEU) consists of system of pulleys, suspensions, belts for supporting and elastic cords. UEU is based on the concept of unloading the body against gravity and to perform movement of weak part of the body. Therapist's hands are free to provide adequate support as required by the patient during exercise training Universal exercise unit, therapy sessions extended are from three to four hours Children and adults have neurological conditions can used. Spider cage is made of metal could be depending on population pediatric or adults. Elastic resistance of cords used to increase strengthen of muscle
  Interventions: Device: universal exercis unit
- effect of functional electrical stimulation on genu recurvatum in diplegic cerbral palsy children (Active Comparator): Functional electrical stimulation (FES) is defined as the electrical stimulation of muscles that have impaired motor control to produce a contraction to obtain functional useful movement
  Interventions: Device: functional electrical stimulation

INTERVENTIONS:
Device: universal exercis unit — Universal exercise unit (UEU) consists of system of pulleys, suspensions, belts for supporting and elastic cords. UEU is based on the concept of unloading the body against gravity and to perform movement of weak part of the body. Therapist's hands are free to provide adequate support as required by the patient during exercise training Universal exercise unit, therapy sessions extended are from three to four hours Children and adults have neurological conditions can used. Spider cage is made of metal could be depending on population pediatric or adults. Elastic resistance of cords used to increase strengthen of muscle
  Arms: effect of universal exercis unit on genu recurvatum in diplegic cerbral palsy children
Device: functional electrical stimulation — Functional electrical stimulation (FES) is defined as the electrical stimulation of muscles that have impaired motor control to produce a contraction to obtain functional useful movement
  Arms: effect of functional electrical stimulation on genu recurvatum in diplegic cerbral palsy children

SUMMARY:
Summary:

Inclusion Criteria:

* Children aged four to eight years.
* Grade of spasticity ranging from 1 to 1+ on the Modified Ashworth scale.
* Classified as Level I or II on the Gross Motor Functional Classification System (GMFCS).
* Ability to follow verbal commands and instructions.

Exclusion Criteria:

* Previous neurological or orthopedic surgery in the lower extremities.
* Botox injection in the lower extremities within the past six months.
* Fixed deformity in the joints of the lower limb.
* Genu recarvatum secondary to surgery.
* Severe hearing and visual defects.

Materials for Subject Selection and Evaluation:

* Modified Ashworth Scale for muscle tone assessment.
* Gross Motor Functional Classification System (GMFCS) for functional activity classification.
* Digital goniometer for measuring the angle of knee hyperextension.
* Lafayette Manual Muscle Tester for quantifying muscle strength.

Methods:

* Assessment of muscle tone using the Modified Ashworth Scale, evaluating spasticity in calf muscles and hip/knee extensors.
* Evaluation of gross motor function using the GMFCS.
* Assessment of genu recarvatum using a digital goniometer.
* Assessment of muscle strength using the Lafayette Manual Muscle Tester, focusing on hamstrings and tibialis anterior muscles.
* Assessment of range of motion in the knee joint using Kinovea software.
* Treatment procedures involving physical therapy sessions with a combination of exercises and interventions tailored to each group (Group A and Group B).

Group A Treatment:

- Designed physical therapy program combined with pulley therapy for muscle strengthening.

Group B Treatment:

- Designed physical therapy program combined with functional electrical stimulation during walking on a treadmill for muscle stimulation.

The interventions in both groups aim to improve muscle strength, range of motion, and functional abilities in children with cerebral palsy.

DETAILED DESCRIPTION:
B)For assessment:

1. Assessment of muscle strength

   * In this study, Lafayette manual muscle tester device will be used to assess muscle strength of hamstrings and tibialis anterior muscles.
   * Test procedures will be demonstrated to each child.
   * For both tests each child will perform three corrected trials and the average will be taken in analysis.

   For tibialis anterior muscle:

   Each child will be lied supine with feet relaxed on the plinth. Hips knees will be in extension and neutral rotation. Each child will be stabilized by straps at pelvis and just above knees, then the examiner will place the device in his hand and put it on the dorsum aspect of examined foot over the metatarsal heads and ask the child to take his/her foot toward him the device

   For hamstrings muscle:

   Each child will be seated with hips and knees flexed 90°. Each child will be stabilized at trunk, pelvis and unexamined limb by straps to prevent any substitutions. The examined limb will be stabilized above examiner hand and in the other hand Lafayette device will be placed. The device will be placed on the posterior lower part of the examined leg then the examiner will ask the child to move his/her lower leg backward against device.
2. Assessment of range of motion in knee joint

   * Using kinovea, Kinovea is a free 2D motion analysis software that enables the establishment of kinematics parameters. This low-cost technology has been used in sports sciences, as well as clinical field and research work. Kinovea is a free, reliable tool that produces valid data, providing an acceptable level of accuracy in angular and linear measurements obtained via digitization of x- and y axis coordinates -Treatment procedures: - •Each child of both group A&B received a designed physical therapy program, attending three sessions per week for three consecutive months. The program used a combination of open-and closed-chain exercises. Exercises for facilitating standing and balance as kneeling and half kneeling exercises, step standing, single limb support, from supine to stand, from prone to stand and standing on balance board, abdominal and core stability exercise on wedge, exercises for strengthening of hamstring and tibialis anterior muscles by using free weights and gait training including walking in stepper between parallel bars and ascending and descending stairs for one hour

     1. Group A Each child in the group A received the designed program physical therapy in addition to pulley therapy, attending three sessions per week for three consecutive months. The duration of the session was one hour that was divided into half an hour for the designed physical therapy program and half an hour for the pull therapy. The pulley therapy is used to strength hamstring and tibialis anterior muscles. The weight used in training is determined by using the one repetition maximum method (I-RM). The 1-RM was taken as the maximum resistance that could be lifted throughout the full ROM. To assess 1-RM, estimate the starting weight to be a little bit less than the child's maximum capacity for lifting. Then for exercises, weight increased gradually in each attempt till the child reached maximum lifting capacity. The added weight ranged from 1 to 5 kg according to the evaluated muscle group. With periods of rest from 1 to 5 minutes allowed before attempting a lift at the next heavier weight. Children performed a mild to moderate load (about 60% 1-RM) for 1 to 2 sets with 8-15 repetitions. For hamstring muscle: each child lied prone on the table inside spider cage. The child stabilized by straps at pelvis and unaffected limb. The affected limb was stabilized at thigh level with lower leg free to move. A band around lower leg attached to upper part of the cage by a rope at foot side. At the end of the rope there was a weight to pull Each child was asked to pull his leg toward him against weight doing one set of 10 repetitions at first up to 1-2 sets of 8-15 repetitions.

        For tibialis anterior: each child lied supine on the table inside spider cage. The child stabilized by straps at pelvis and unaffected limb. The affected limb was stabilized by straps at thigh and lower leg with foot free to move. A band around foot attached to upper part of the cage by a rope at foot side. At the end of the rope there was a weight to pull. Each child was asked to pull his foot toward him against weight doing one set of 10 repetitions up to 1-2 sets of 8-15 repetitions for 20 minutes.
     2. Group B Each child in group B receive the designed program plus the functional electrical stimulation for 30minutes on hamstring muscle and tibalis anterior muscle during walking on tread-mail with the following parameters: - Pulse frequency 25-40 HZ, pulse duration 250 to 300 msec with on: off time 1:2 for 20 minutes electrodes will attach to peroneal (at the back of the fibular head) and the tibalis anterior muscle (5 cm below the fibular head) and then adjust to create ankle dorsiflexion with avoiding the inversion.

A pair of electrodes stimulated the hamstring muscle near the motor on the motor point on both muscle of bices femoris, semitendinosus and semimembranosus with avoiding the rotation.

ELIGIBILITY:
Inclusion Criteria:

1. Their age will be ranged from four to eight years.
2. Their grade of spasticity will be from 1 to 1+ according to Modified Ashworth scale
3. They will be on Level I and II according to Gross Motor Functional Classification System (GMFCS)
4. The child will be able to follow verbal commands and instructions.

Exclusion Criteria:

- The children will be excluded if they have one of the following:

1. Previous neurological or orthopedic surgery in the lower extremities.
2. Botox injection in the lower extremities in the past 6 months. 4-Fixed deformity in the joints of lower limb.

5- Genu recarvatum secondary to surgery 6- Severe hearing and visual defect.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
muscle strength using muscle tester device | 3 months
  Muscle strength can be measured by estimating a person's one repetition maximum (1RM) - a measurement of the greatest load (in kg) that can be fully moved (lifted, pushed, or pulled) once without failure
  -For both tests each child will perform three corrected trials and the average will be taken in analysis
Range of motion using kinoviea software and digital goniometer | 3 months
  - Kinovea is a free 2D motion analysis software that enables the establishment of kinematics parameters. This low-cost technology has been used in sports sciences, as well as clinical field and research work. Kinovea is a free, reliable tool that produces valid data, providing an acceptable level of accuracy in angular and linear measurements obtained via digitization of x- and y axis coordinates an angle measured in degrees (°)through which a joint moves away from a reference position
range of motion for the joint using digital geniometer | 3 months
  measure the angle of the joint by degree (°)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud R Elsharkawy, bachelor, Principal Investigator — Demonstrator of physical therapy at Alsalam university; Abd Elaziz Ali sherif, PHD, Study Chair — professor of pediatric department Faculty of physical therapy; Osama Abd Elfattah El-Agamy, PHD, Study Chair — Professor and head of department of pediatric faculty of medicine; Sara Y Abdel Elglil Elsebahy, Study Director — Lecturer of pediatric department Faculty of physical therapy
Locations (1):
- Physical Therapy, Kafr ash Shaykh, Egypt

REFERENCES:
- [Derived] Elsharkawy MR, Sherif AEA, Sarhan EE, El-Agamy OA, Elsebahy SY. Effect of Universal Exercise Unit Versus Functional Electrical Stimulation on Genu Recurvatum in Diplegic Cerebral Palsy Children. J Musculoskelet Neuronal Interact. 2025 Mar 1;25(1):109-118. doi: 10.22540/JMNI-25-109. PMID 40024234